CLINICAL TRIAL: NCT03035487
Title: Urology of Virginia Case Series
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Exact Imaging (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 2016-UHR-001
Record Dates: First submitted 2017-01-16; First posted 2017-01-30 (Estimated); Results first posted 2019-03-04 (Actual); Last update posted 2019-05-15 (Actual); Status verified 2019-04

CONDITIONS: Prostate Cancer; Cancer of the PROSTATE; Prostatic Neoplasm
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Micro-ultrasound (Experimental): Transrectal micro-ultrasound guided prostate biopsy, where images will be compared with images from standard of care modalities:
  * Low resolution transrectal ultrasound examination ("LR-TRUS")
  * Multi-parametric MRI ("mpMRI") examination performed according to the PI-RADS v2 protocol
  Interventions: Device: Ultrasound guided prostate exam using SOC ultrasound system; Device: mpMRI guided prostate examination using PI-RADS v2; Device: High-resolution micro-ultrasound guided prostate biopsy

INTERVENTIONS:
Device: Ultrasound guided prostate exam using SOC ultrasound system
Device: mpMRI guided prostate examination using PI-RADS v2 — mpMRI guided prostate examination using standard of care MRI system
Device: High-resolution micro-ultrasound guided prostate biopsy
  Other Names: ExactVu micro-ultrasound imaging system

SUMMARY:
The investigational protocol describes a small case series designed to compare three imaging modalities for use in visualizing prostate cancer.

The three modalities to be tested are: transrectal micro-ultrasound , and conventional resolution transrectal ultrasound (LR-TRUS) (both as implemented on ExactVu, the multi-frequency novel micro-ultrasound system under investigation), and multi-parametric MRI (mpMRI).

These modalities will be used for guiding systematic (standard, random, extended sextant) plus image-guided targeted prostate biopsies among men with known cancer and an indication for prostate biopsy.

In the case of mpMRI, biopsy will be performed under micro-ultrasound guidance with the radiology report used for targeting.

DETAILED DESCRIPTION:
This trial will enroll nine men with an indication for a prostate biopsy.

The primary objective of the study is to provide guidance to clinicians who will be using the ExactVu system on the appearance of suspicious foci, and the difference between the appearance of these foci in LR-TRUS, mpMRI and transrectal micro-ultrasound images.

The study is being conducted based on the hypothesis that a series of same-subject comparisons will clearly demonstrate the differences in appearance between the modalities.

Procedures in the study are:

* obtain informed consent for the subject
* image the subject using mpMRI according to the PI-RADS v2 protocol, and obtain radiologist's report
* perform biopsy procedure using micro-ultrasound (this may be conducted in a separate subject visit)
* prepare biopsy specimens for pathology
* record all procedure details in a case report form, including pathology and mpMRI reports

The primary endpoint will be a standardized description using keywords of each biopsy sample region. These descriptions will be recorded during the blinded readings after the procedure to avoid added procedure time and will be used to compare appearance between the modalities.

Secondary endpoints are the pathological result of each biopsy sample (Gleason Score and percentage of cancer in sample), and risk score identified on imaging. Both of these values are per-sample, with 12 systematic samples per subject plus any additional targeted samples warranted by standard of care.

ELIGIBILITY:
Inclusion Criteria:

1. All men ≥ 40 years age and <80 years of age with a history of prostate cancer and an indication for a prostate biopsy will be offered inclusion in the study. Typical indications for biopsy include abnormal PSA (prostate specific antigen) and/or abnormal DRE (digital rectal exam) and/or history of prostate cancer.
2. PSA<50
3. Clinical stage < cT2c

Exclusion Criteria:

Patients will be excluded from being included in the investigation if any of the following is true:

1. Men undergoing TRUS-guided prostate biopsy in the OR under anesthesia
2. Men with known prostate volume (from prior imaging) of > 60cc
3. Men with anorectal abnormalities preventing TRUS-guided prostate biopsy
4. Men who are unable to provide their own informed consent
5. Men who have contraindications to MRI or gadolinium chelate contrast

Ages: 40 Years to 79 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2016-12; Primary Completion 2016-12 (Actual); Study Completion 2018-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Urology of Virginia, Virginia Beach, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Micro-ultrasound: Transrectal micro-ultrasound guided prostate biopsy, where images will be compared with images from standard of care modalities:
  * Low resolution transrectal ultrasound examination ("LR-TRUS")
  * Multi-parametric MRI ("mpMRI") examination performed according to the PI-RADS v2 protocol
  Ultrasound guided prostate exam using SOC ultrasound system
  mpMRI guided prostate examination using PI-RADS v2: mpMRI guided prostate examination using standard of care MRI system
  High-resolution micro-ultrasound guided prostate biopsy
Period: Overall Study
Arm/Group | Micro-ultrasound
Started | 9
Completed | 9
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Micro-ultrasound
Number analyzed (Participants) | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 9
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 9

OUTCOME MEASURES:

1. Primary Outcome: Keyword Description of Each Biopsy Sample
Description: The primary endpoint will be a standardized description using keywords of each biopsy sample region. These descriptions will be recorded during the blinded readings after the procedure to avoid added procedure time and will be used to compare appearance between the modalities. Keywords will be derived from standard lexicons such as PI-RADS for MRI and PRI-MUS for Micro-Ultrasound.
Time Frame: For each patient, keywords will be assigned within one week following the patient's procedure.
Measure: Number; unit: percentage significant cancers detected
Arm/Group | Micro-ultrasound
Number analyzed (Participants) | 9
percentage significant cancers detected | 89

ADVERSE EVENTS:
Arm/Group | Micro-ultrasound
Serious Adverse Events (participants affected / at risk) | 0/9
Other Adverse Events (participants affected / at risk) | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No